CLINICAL TRIAL: NCT01849783
Title: Single Autologous Transplant Followed by Consolidation and Maintenance for Participants ≥ 65 Years of Age Diagnosed With Multiple Myeloma or a Related Plasma Cell Malignancy
Brief Title: Autologous Stem Cell Transplant Followed By Maintenance Therapy in Treating Elderly Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Margarida Magalhaes-Silverman (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Margarida Magalhaes-Silverman, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201208775; 10120146; P30CA086862 (NIH); NCI-2013-00883 (Other: NCI CTRP)
Record Dates: First submitted 2013-05-06; First posted 2013-05-09 (Estimated); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Extramedullary Plasmacytoma; Isolated Plasmacytoma of Bone; Light Chain Deposition Disease; Primary Systemic Amyloidosis; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; Cisplatin; Doxorubicin; Cyclophosphamide; Etoposide; Bortezomib; Thalidomide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- autologous stem cell transplant (Experimental): Induction : DPACE(dexamethasone,cisplatin,doxorubicin,cyclophosphamide,etoposide) chemotherapy plus stem cell collection. Additional stem cell collection and/or chemotherapy may be required.
  After collection, participants will receive dexamethasone x 4 days every 14 days.
  Transplant: The transplant preparative regimen will be bortezomib/thalidomide/dexamethasone/melphalan.
  Once recovered, participants start thalidomide daily and dexamethasone x 4 days every 21 days.
  Consolidation (if administered): VDT-PACE(bortezomib,dexamethasone,thalidomide,cisplatin,doxorubicin,cyclophosphamide, etoposide)
  Maintenance: Year 1 - VTD (bortezomib, thalidomide, dexamethasone) cycles. Year 2 - VCD (bortezomib, cyclophosphamide, dexamethasone)cycles.
  Interventions: Drug: dexamethasone; Drug: cisplatin; Drug: doxorubicin; Drug: cyclophosphamide; Drug: etoposide; Drug: bortezomib; Drug: thalidomide; Drug: melphalan; Procedure: autologous stem cell transplant

INTERVENTIONS:
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: doxorubicin — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given IV or PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: thalidomide — Given PO
  Other Names: Kevadon; Synovir; THAL; Thalomid
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Procedure: autologous stem cell transplant

SUMMARY:
This phase II trial investigates whether patients greater than or equal to 65 years of age diagnosed with myeloma or another plasma cell malignancy will have better outcomes with transplant followed by maintenance therapy, as primarily measured by progression-free survival, versus non-transplant approaches.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression-free survival (PFS) from the start of dexamethasone, cisplatin, Adriamycin (doxorubicin),Cytoxan (cyclophosphamide), etoposide (DPACE) for all participants who have had at least one day of protocol treatment.

II. To evaluate how well such therapy is tolerated in patients mainly over the age of 65 years by assessing severe complications (intensive care unit [ICU] admission, death) and the percentage of participants able to complete the full course of therapy.

SECONDARY OBJECTIVES:

I. To evaluate Quality-Of-Life post-transplant using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire QLQ-C30 and QLC-MY20.

OUTLINE:

INDUCTION THERAPY: Patients receive dexamethasone orally (PO) on days 1-4 and 8-11, cisplatin intravenously (IV) continuously, doxorubicin hydrochloride IV continuously, cyclophosphamide IV, and etoposide IV on days 1-4. Patients then receive pegfilgrastim subcutaneously (SQ) on days 6 and 13 and undergo collection of stem cells when white blood cell (WBC) and cluster of differentiation (CD)34 counts are within program range. Following stem cell collection, patients may receive interim dexamethasone PO on days 1-4, every 14 days at the discretion of the treating physician.

TRANSPLANT: Beginning between 4 weeks to 6 months after the first day of induction therapy, patients receive as transplant conditioning regimen dexamethasone PO on days -4 to -1 and days +2 through +5, bortezomib IV bolus on days -4, -1, 2, and 5, thalidomide PO on days -4 to 5, and melphalan IV on days -4 and -1. Patients undergo autologous peripheral blood stem cell transplant (PBSCT) on day 0. Between transplant and consolidation therapy, patients receive dexamethasone PO on days 1-4 every 21 days and thalidomide PO daily.

CONSOLIDATION THERAPY: If administered, post-transplant consolidation may begin 4-6 weeks after transplant but should occur no more than 4 months later. Most patients will not receive consolidation. Those that do will receive dexamethasone PO on days 1-4 and 8-11, thalidomide PO on days 1-11, bortezomib IV on days 1, 4, 8, and 11, cisplatin IV continuously, doxorubicin hydrochloride IV continuously, cyclophosphamide IV continuously, and etoposide IV continuously on days 1-4.

MAINTENANCE THERAPY YEAR 1: Beginning 6 weeks-6 months after consolidation therapy or 4 weeks to 6 months after transplant if consolidation is skipped, patients receive bortezomib IV bolus on days 1, 4, 15, and 18, thalidomide PO QD on days 1-28, and dexamethasone PO on days 1-4 and 15-18. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY YEAR 2: Patients receive bortezomib IV on days 1, 4, 15, and 18, cyclophosphamide PO or IV on days 1 and 15, and dexamethasone PO QD on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at least once annually at the study center, but serum for MM marker results will be sent to the study site for close monitoring of PFS .

ELIGIBILITY:
Inclusion Criteria:

* Participants must have had a diagnosis of symptomatic multiple myeloma (MM), MM + amyloidosis, or POEMS (osteosclerotic myeloma: polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes) requiring treatment; participants with a previous history of smoldering myeloma will be eligible if there is evidence of progressive disease requiring chemotherapy; Note that study participants do not need to have active disease at the time of study entry, as participants may have received up to 12 months of prior chemotherapy, which might have induced a response
* Protein criteria must be present at diagnosis (quantifiable M-component of IgG, IgA, IgD, or IgE and/or urinary kappa or lambda light chain, Bence-Jones protein, or Free Kappa Light Chain or Free Lambda Light Chain) in order to evaluate response. Non-secretory participants are eligible provided the participant has > 20% plasmacytosis OR multiple (≥3) plasmacytomas or lesions on MRI at the time of diagnosis or study enrollment , OR the presence of lesions on PET/CT scan or skeletal survey at diagnosis or study enrollment.
* Participants must have received ≤12 months of prior chemotherapy for this disease without evidence of progressive disease with treatment. Participants may have received prior radiotherapy provided approval has been obtained from the PI. Participants with a history of radiation who have a platelet count <150,000 due to radiation (disease, chemo, and other factors have been ruled out) will be excluded from this study.
* Participants must not have had a prior transplant
* Participants must be 65-85 years of age at the time of study entry.
* Ejection fraction by echocardiogram (ECHO) or multigated acquisition scan (MUGA) of >= 40% performed
* Participants must have adequate pulmonary function studies (PFTs), >= 50% of predicted on mechanical aspects (forced expiratory volume in 1 second [FEV^1}, forced vital capacity [FVC]) and diffusion capacity (diffusion capacity of the lung for carbon monoxide [DLCO]) >= 50% of predicted (adjusted for hemoglobin); if the participant is unable to complete pulmonary function tests (PFTs) due to disease-related pain or other circumstances that make it difficult to reliably perform PFTs, documentation of pulmonary function adequate for transplant will occur via a CT scan without evidence of major pulmonary disease, and arterial blood gas results
* Participants must have a creatinine < 3 mg/dl and a GFR >30mL/min/1.73m2
* Participants must have a performance status of 0-2 based on Eastern Cooperative Oncology Group (ECOG) criteria; participants with a poor performance status (3-4) based solely on bone pain will be eligible, provided there is documentation to verify this
* Participants must sign the most current institutional review board (IRB)-approved study (informed consent form) ICF

Exclusion Criteria:

* Prior autologous or allogeneic transplant
* Progressive disease on prior treatment
* Platelet count < 30 x 10^9/L, unless myeloma-related; if MM-related (hypercellular marrow biopsy of > 80% and packed with at least 80% plasma cells) the enrolling investigator must document this
* > Grade 3 neuropathy
* Known hypersensitivity to bortezomib, boron, or mannitol
* Uncontrolled diabetes on appropriate therapy
* Recent (=< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension on appropriate therapy, or difficult-to-control cardiac arrhythmias
* Participants must not have a creatinine >3 mg/dl or a GFR <30mL/min/1.73m2.
* Participants must not have a concurrent malignancy unless it can be adequately treated by non-chemotherapeutic intervention; participants may have a history of prior malignancy, provided that he/she has not had any chemotherapy within 365 days of study entry AND that life expectancy exceeds 5 years at the time of study entry
* Participants must not have life-threatening co-morbidities

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margarida Magalhaes-Silverman, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Autologous Stem Cell Transplant: Induction : DPACE(dexamethasone,cisplatin,doxorubicin,cyclophosphamide,etoposide) chemotherapy plus stem cell collection. Additional stem cell collection and/or chemotherapy may be required.
  After collection, participants will receive dexamethasone x 4 days every 14 days.
  Transplant: The transplant preparative regimen will be bortezomib/thalidomide/dexamethasone/melphalan.
  Once recovered, participants start thalidomide daily and dexamethasone x 4 days every 21 days.
  Consolidation (if administered): VDT-PACE(bortezomib,dexamethasone,thalidomide,cisplatin,doxorubicin,cyclophosphamide, etoposide)
  Maintenance: Year 1 - VTD (bortezomib, thalidomide, dexamethasone) cycles. Year 2 - VCD (bortezomib, cyclophosphamide, dexamethasone)cycles.
  dexamethasone: Given PO
  cisplatin: Given IV
  doxorubicin: Given IV
  cyclophosphamide: Given IV or PO
  etoposide: Given IV
  bortezomib: Given IV
  thalidomide: Given PO
  melphalan: Given IV
  autologous stem cell transplant
Period: Overall Study
Arm/Group | Autologous Stem Cell Transplant
Started | 41
Completed | 19
Not Completed | 22
Not completed — Adverse Event | 5
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Unable to comply | 2
Not completed — Disease progression | 11

BASELINE CHARACTERISTICS:
Arm/Group | Autologous Stem Cell Transplant
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 41
Age, Continuous [Mean (Full Range); unit: years] | 69 [65 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 38
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (mPFS)
Description: PFS is defined as the time from the start of DPACE to the date of first documentation of disease progression as assessed by the International Myeloma Working Group response criteria or death due to any cause. Progression is defined using the International Myeloma Working Group response criteria, an increase of greater than or equal to 25% from the lower response value.
Time Frame: From the start of DPACE for all participants who have had at least one day of protocol treatment. Up to 6 years.
Population: Participants who have had at least one day of protocol treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Autologous Stem Cell Transplant
Number analyzed (Participants) | 41
months | 76.4 [43.6 to NA] — 1-sided 95% confidence interval reported. Study designed to test whether regimen would increase PFS using 1-sided test at 5% significance level. In accordance with statistical hypothesis,1-sided 95% confidence interval is reported. The form does not provide option for 1-sided confidence interval; only options for 2-sided confidence intervals. Since a 1-sided confidence interval only has 1 bound, NA entered for the upper bound because there is no upper bound.

2. Primary Outcome: Percentage of Participants With Serious Treatment-Related Complications
Description: Percentage of participants with severe complications defined at ICU admission and death, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.
Time Frame: From the start of DPACE for all participants who have had at least one day of protocol treatment. Up to 6 years.
Population: Participants who have had at least one day of protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous Stem Cell Transplant
Number analyzed (Participants) | 41
Participants | 4

3. Primary Outcome: Percentage of Participants Able to Complete Full Course Therapy
Description: Percentage of participants able to complete the full course of therapy.
Time Frame: Up to 6 years
Population: Participants who received at least one day of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous Stem Cell Transplant
Number analyzed (Participants) | 41
Participants | 24

4. Secondary Outcome: Mean Change in Quality-Of-Life Indicators Post-Transplant
Description: Measured using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) and Multiple Myeloma module (QLQ-MY20). The EORTC QLQ-C30 includes functional scales (physical, role, emotional, cognitive, and social) and global health status. The EORTC QLQ-MY20 includes disease symptoms and treatment side effects scales. Scores are averaged and transformed to 0-100 scale. For functional and global health status, a positive change from baseline (pre-DPACE) indicates improvement whereas for the symptom scales a negative change from baseline (pre-DPACE) indicates improvement.
Time Frame: Pre-DPACE, Pre-maintenance, every 6 months for up to 2 years during maintenance. Up to 6 years.
Population: Participants who received at least one day of study treatment. Globally, there were 37 patients who were included in at least one of the estimated mean change scores being reported. Four patients were not included due to not completing the baseline questionnaire making it impossible to calculate change from baseline (n=3) or did not complete the questionnaire at any time point (n=1).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Autologous Stem Cell Transplant
Number analyzed (Participants) | 37
score on a scale
  Change in Physical Functioning at Pre-Maintenance: number analyzed (Participants) | 30
  Change in Physical Functioning at Pre-Maintenance | 1.3 [-5.2 to 7.9]
  Change in Physical Functioning at Maintenance Cycle 6: number analyzed (Participants) | 31
  Change in Physical Functioning at Maintenance Cycle 6 | -0.6 [-7.1 to 5.9]
  Change in Physical Functioning at Maintenance Cycle 12: number analyzed (Participants) | 26
  Change in Physical Functioning at Maintenance Cycle 12 | 1.1 [-5.6 to 7.8]
  Change in Physical Functioning at Maintenance Cycle 18: number analyzed (Participants) | 24
  Change in Physical Functioning at Maintenance Cycle 18 | 5.4 [-1.5 to 12.3]
  Change in Physical Functioning at Maintenance Cycle 24: number analyzed (Participants) | 22
  Change in Physical Functioning at Maintenance Cycle 24 | 4.6 [-2.6 to 11.7]
  Change in Role Functioning at Pre-Maintenance: number analyzed (Participants) | 28
  Change in Role Functioning at Pre-Maintenance | 7.4 [-5.5 to 20.4]
  Change in Role Functioning at Maintenance Cycle 6: number analyzed (Participants) | 30
  Change in Role Functioning at Maintenance Cycle 6 | 8.7 [-4.0 to 21.5]
  Change in Role Functioning at Maintenance Cycle 12: number analyzed (Participants) | 26
  Change in Role Functioning at Maintenance Cycle 12 | 4.4 [-8.7 to 17.5]
  Change in Role Functioning at Maintenance Cycle 18: number analyzed (Participants) | 23
  Change in Role Functioning at Maintenance Cycle 18 | 7.0 [-6.6 to 20.5]
  Change in Role Functioning at Maintenance Cycle 24: number analyzed (Participants) | 22
  Change in Role Functioning at Maintenance Cycle 24 | 6.0 [-8.0 to 20.0]
  Change in Emotional Functioning at Pre-Maintenance: number analyzed (Participants) | 31
  Change in Emotional Functioning at Pre-Maintenance | 8.7 [2.5 to 14.9]
  Change in Emotional Functioning at Maintenance Cycle 6: number analyzed (Participants) | 32
  Change in Emotional Functioning at Maintenance Cycle 6 | 5.5 [-0.6 to 11.6]
  Change in Emotional Functioning at Maintenance Cycle 12: number analyzed (Participants) | 28
  Change in Emotional Functioning at Maintenance Cycle 12 | 1.4 [-4.9 to 7.7]
  Change in Emotional Functioning at Maintenance Cycle 18: number analyzed (Participants) | 24
  Change in Emotional Functioning at Maintenance Cycle 18 | 5.8 [-1.0 to 12.5]
  Change in Emotional Functioning at Maintenance Cycle 24: number analyzed (Participants) | 24
  Change in Emotional Functioning at Maintenance Cycle 24 | 8.3 [1.3 to 15.2]
  Change in Cognitive Functioning at Pre-Maintenance: number analyzed (Participants) | 31
  Change in Cognitive Functioning at Pre-Maintenance | 0.4 [-7.1 to 7.9]
  Change in Cognitive Functioning at Maintenance Cycle 6: number analyzed (Participants) | 31
  Change in Cognitive Functioning at Maintenance Cycle 6 | -4.6 [-12.0 to 2.9]
  Change in Cognitive Functioning at Maintenance Cycle 12: number analyzed (Participants) | 28
  Change in Cognitive Functioning at Maintenance Cycle 12 | -5.1 [-12.8 to 2.5]
  Change in Cognitive Functioning at Maintenance Cycle 18: number analyzed (Participants) | 25
  Change in Cognitive Functioning at Maintenance Cycle 18 | -6.0 [-14.0 to 2.1]
  Change in Cognitive Functioning at Maintenance Cycle 24: number analyzed (Participants) | 24
  Change in Cognitive Functioning at Maintenance Cycle 24 | -3.6 [-11.9 to 4.7]
  Change in Social Functioning at Pre-Maintenance: number analyzed (Participants) | 30
  Change in Social Functioning at Pre-Maintenance | -1.0 [-11.0 to 9.1]
  Change in Social Functioning at Maintenance Cycle 6: number analyzed (Participants) | 31
  Change in Social Functioning at Maintenance Cycle 6 | 2.7 [-7.2 to 12.6]
  Change in Social Functioning at Maintenance Cycle 12: number analyzed (Participants) | 25
  Change in Social Functioning at Maintenance Cycle 12 | -4.9 [-15.3 to 5.6]
  Change in Social Functioning at Maintenance Cycle 18: number analyzed (Participants) | 24
  Change in Social Functioning at Maintenance Cycle 18 | 0.8 [-9.9 to 11.6]
  Change in Social Functioning at Maintenance Cycle 24: number analyzed (Participants) | 23
  Change in Social Functioning at Maintenance Cycle 24 | -1.5 [-12.7 to 9.7]
  Change in Global Health Status at Pre-Maintenance: number analyzed (Participants) | 31
  Change in Global Health Status at Pre-Maintenance | 5.4 [-2.7 to 13.5]
  Change in Global Health Status at Maintenance Cycle 6: number analyzed (Participants) | 32
  Change in Global Health Status at Maintenance Cycle 6 | 0.2 [-7.8 to 8.3]
  Change in Global Health Status at Maintenance Cycle 12: number analyzed (Participants) | 28
  Change in Global Health Status at Maintenance Cycle 12 | -3.1 [-11.4 to 5.1]
  Change in Global Health Status at Maintenance Cycle 18: number analyzed (Participants) | 25
  Change in Global Health Status at Maintenance Cycle 18 | -0.1 [-8.8 to 8.5]
  Change in Global Health Status at Maintenance Cycle 24: number analyzed (Participants) | 24
  Change in Global Health Status at Maintenance Cycle 24 | 3.4 [-5.6 to 12.3]
  Change in Distress Symptoms at Pre-Maintenance: number analyzed (Participants) | 32
  Change in Distress Symptoms at Pre-Maintenance | 6.2 [1.2 to 11.2]
  Change in Distress Symptoms at Maintenance Cycle 6: number analyzed (Participants) | 32
  Change in Distress Symptoms at Maintenance Cycle 6 | 5.9 [0.9 to 10.8]
  Change in Distress Symptoms at Maintenance Cycle 12: number analyzed (Participants) | 28
  Change in Distress Symptoms at Maintenance Cycle 12 | 5.7 [0.5 to 10.9]
  Change in Distress Symptoms at Maintenance Cycle 18: number analyzed (Participants) | 25
  Change in Distress Symptoms at Maintenance Cycle 18 | 3.8 [-1.7 to 9.3]
  Change in Distress Symptoms at Maintenance Cycle 24: number analyzed (Participants) | 24
  Change in Distress Symptoms at Maintenance Cycle 24 | 5.3 [-0.4 to 11.0]
  Change in Side Effects of Treatment at Pre-Maintenance: number analyzed (Participants) | 32
  Change in Side Effects of Treatment at Pre-Maintenance | -3.3 [-8.0 to 1.3]
  Change in Side Effects of Treatment at Maintenance Cycle 6: number analyzed (Participants) | 32
  Change in Side Effects of Treatment at Maintenance Cycle 6 | -0.7 [-5.3 to 3.9]
  Change in Side Effects of Treatment at Maintenance Cycle 12: number analyzed (Participants) | 28
  Change in Side Effects of Treatment at Maintenance Cycle 12 | -5.1 [-9.8 to -0.3]
  Change in Side Effects of Treatment at Maintenance Cycle 18: number analyzed (Participants) | 25
  Change in Side Effects of Treatment at Maintenance Cycle 18 | -2.4 [-7.4 to 2.5]
  Change in Side Effects of Treatment at Maintenance Cycle 24: number analyzed (Participants) | 24
  Change in Side Effects of Treatment at Maintenance Cycle 24 | -2.7 [-7.8 to 2.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected pre-study, post-induction, pre-transplant, pre-consolidation, during maintenance therapy and long term follow-up. Up to 6 years overall.
Description: Adverse events (AEs ≥ grade 3) were recorded. AEs were not recorded by start and stop date but by phase of treatment in which the AE occurred. AEs will be recorded as the worst grade achieved during that phase of treatment.
Groups:
- D-PACE/Induction: Initial chemotherapy will consist of 1 cycle of combination D-PACE chemotherapy and peripheral blood stem cell collection.
- Post D-PACE/Pre-Transplant: Following D-PACE and Peripheral Blood Stem Cell (PBSC) collection, participants may receive interim dexamethasone at 20mg days 1-4 every 14 days, but this may be omitted by the treating physician
- Transplant: Transplant should preferably occur 6 weeks after the induction PACE continuous infusion has been completed, but can occur as early as 4 weeks and as late as 3 months if the participant fails to mobilize stem cells after the PACE administration
- Post-transplant/Consolidation: Participants will receive dexamethasone 20 mg oral days 1-4 every 21 days and thalidomide 100 mg oral and daily in the interim between transplant and consolidation.
  If administered, post-transplant consolidation therapy should begin 4-6 weeks after transplant, but should occur no later than 4 months after transplant. Consolidation will consist of one cycle of VDT-PACE.
- Maintenance Therapy, Year 1; Maintenance Therapy, Year 2: Maintenance will begin 4 weeks to 6 months after transplant, or between 6 weeks to 6 months after consolidation if administered. This is considered standard of care
- Long Term Follow-up: Study participants will be evaluated at the study center at least once per year.
Arm/Group | D-PACE/Induction | Post D-PACE/Pre-Transplant | Transplant | Post-transplant/Consolidation | Maintenance Therapy, Year 1 | Maintenance Therapy, Year 2 | Long Term Follow-up
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 1/39 | 0/38 | 1/37 | 0/31 | 0/24
Serious Adverse Events (participants affected / at risk) | 14/41 | 2/41 | 8/39 | 4/38 | 11/37 | 9/31 | 1/24
Other Adverse Events (participants affected / at risk) | 41/41 | 8/41 | 38/39 | 8/38 | 27/37 | 22/31 | 3/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-PACE/Induction (N=41) | Post D-PACE/Pre-Transplant (N=41) | Transplant (N=39) | Post-transplant/Consolidation (N=38) | Maintenance Therapy, Year 1 (N=37) | Maintenance Therapy, Year 2 (N=31) | Long Term Follow-up (N=24)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-PACE/Induction (N=41) | Post D-PACE/Pre-Transplant (N=41) | Transplant (N=39) | Post-transplant/Consolidation (N=38) | Maintenance Therapy, Year 1 (N=37) | Maintenance Therapy, Year 2 (N=31) | Long Term Follow-up (N=24)
Anemia (Blood and lymphatic system disorders) | 15 (15) | 2 (2) | 30 (33) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
Corneal ulcer (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (8) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 6 (6) | 3 (4) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 2 (2) | 7 (7) | 1 (1) | 6 (6) | 23 (47) | 14 (19) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 41 (42) | 8 (8) | 36 (36) | 8 (10) | 27 (113) | 22 (85) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 33 (33) | 1 (1) | 31 (31) | 2 (2) | 3 (4) | 3 (3) | 0 (0)
Pancreatic enzymes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 35 (35) | 1 (1) | 38 (39) | 3 (3) | 3 (5) | 5 (10) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 39 (40) | 0 (0) | 38 (38) | 3 (3) | 4 (25) | 4 (4) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 4 (6) | 1 (1) | 4 (24) | 4 (8) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 10 (10) | 1 (1) | 22 (22) | 3 (3) | 11 (20) | 9 (10) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT01849783/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT01849783/ICF_001.pdf